CLINICAL TRIAL: NCT04794231
Title: Comparison of Chlorhexidine Impregnated Dressing and Standard Dressing for the Prevention of Central-line Associated Blood Stream Infection and Colonization in Critically Ill Pediatric Patients: A Randomized Controlled Trial
Brief Title: Comparison of Chlorhexidine Impregnated Dressing and Standard Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Muhterem Duyu, Assistant Proffesor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/0203
Record Dates: First submitted 2021-02-22; First posted 2021-03-12 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Catheter-Related Infections
Keywords: Chlorhexidine dressing; Central venous catheter; Central line associated bloodstream infection; Colonization; Pediatric critical care
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The laboratory microbiologist was blinded to the study groups. The two dressings were visibly different, and consequently, it was not possible to blind the patients, PICU staff or the investigators who collected data in the PICU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dressing group (Active Comparator): Patients were randomly assigned to one of two dressings, both of which were being actively used as part of standard care.
  Interventions: Other: Standard dressing
- Chlorhexidine gluconate -impregnated dressing group (Active Comparator): Patients were randomly assigned to one of two dressings, both of which were being actively used as part of standard care.
  Interventions: Other: Chlorhexidine gluconate -impregnated dressing group

INTERVENTIONS:
Other: Standard dressing — a standard breathable, hypoallergenic, transparent dressing (TegadermTM 1635 [8.5 x 10.5cm] or 1633 [7 × 8.5 cm] depending on patient size; 3M, Neuss, Germany)
  Arms: Standard dressing group
Other: Chlorhexidine gluconate -impregnated dressing group — A chlorhexidine gluconate -gel impregnated transparent dressing (TegadermTM CHG 1660R [7 x 8.5 cm] or [11.5 x 8.5 cm] depending on patient size; 3M, Neuss, Germany).
  Arms: Chlorhexidine gluconate -impregnated dressing group

SUMMARY:
Investigators have designed a single-center randomized controlled trial to compare chlorhexidine gluconate (CHG)-impregnated dressing and standard dressing with respect to their effects on the infection outcomes. The study was condcuted in the pediatric intensive care unit in the 18 months period.

DETAILED DESCRIPTION:
The single-center randomized controlled trial study aimed to compare chlorhexidine gluconate (CHG)-impregnated dressing and standard dressing with respect to their effects on the frequency of central-line associated bloodstream infection (CLABSI), catheter related bloodstream infection (CRBSI), primary bloodstream infection (BSI) and catheter colonization in critically ill pediatric patients with short-term non-tunneled central venous catheter (CVC) in a pediatric intensive care unit (PICU) of a tertiary referral hospital in Turkey.. Pediatric patients aged 1 month to 18 years admitted to our PICU between May 2018 and December 2019, who had received placement of a short-term non-tunneled CVC which had stayed in place for at least 48 hours were included into the study. The patients were grouped with respect to the type of catheter fixation they had received, either with CHG-impregnated dressing or standard dressing, which were assigned in a randomized fashion. The groups were compared with regard to the frequencies of CLABSI, CRBSI, primary BSI and catheter colonization, as well as microorganism etiology. Any adverse event related to catheter dressing were recorded. Independent risk factors of CLABSI frequency were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* being aged age less than 18 years old,
* providing informed consent to participate in the study
* insertion of a short term non-tunneled, percutaneously inserted CVC (jugular, subclavian, or femoral) that would remain in place for greater than 48 hours during PICU admission.

Exclusion Criteria:

Patients were excluded if they:

* had known allergies to CHG-impregnated or standard dressing,
* would receive insertion of any other type of CVC device (e.g., peripherally inserted CVC, tunneled CVC), were included in the study previously,
* had a current BSI (positive blood culture within 48 hours),
* had received CVC insertion within the 30 days prior to PICU admission.

Additionally, investigators also excluded patients in which

* catheterization had not been performed by the PICU specialist,
* those that were discharged from the PICU with indwelling CVC,
* patients who received extracorporeal membrane oxygenation,

Individuals in which the following events were recorded:

* Accidental catheter removal,
* CVC removal before 48 hours, and
* death within 48 hours after CVC insertion.

In the event that a patient required CVC re-insertion after the initial catheter was removed (due to any reason), only the first application was included in the study -given that any other exclusion criteria did not exclude the patient. Finally, if a patient required catheter reinsertion before the completion of the 48-hour catheter-infection monitoring of the initial application, the first catheterization was excluded from the study.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 307 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Catheter-related bloodstream infection rate | Up to 7 days after catheter removal
  Catheter infections were identified according to NHSN and IDSA criteria. Catheter-related bloodstream infection defined as bacteremia/fungemia in a patient with an intravascular catheter with at least 1 positive blood culture obtained from a peripheral vein sampled immediately before or within 48 hours after catheter removal, clinical manifestations of infections (ie, fever, chills, and/or hypotension), and no apparent source for the bloodstream infection except the catheter.
Central-line associated bloodstream infection rate | Up to 7 days after catheter removal
  The presence of either catheter-related bloodstream infections or primary bloodstream infection
Primary bloodstream infection rate | Up to 7 days after catheter removal
  The presence of patients with central venous catheter who had (i) at least one positive blood culture, (ii) clinical manifestation of infection (i.e., fever, chills, and/or hypotension), (iii) no apparent source for the BSI except the catheter, and (iv) no positivity in catheter culture
Catheter colonization rate | Up to 7 days after catheter removal
  The growth of >15 CFU in catheter tip cultures in the absence of local or systemic signs of infection or lack of growth in the two blood samples, or in the event that the two cultures showed growth of the same microorganism which was different from the microorganism isolated in the culture of the catheter tip

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet Üniversitesi Göztepe Eğitim Ve Araştirma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After research will be ended, all data (except personel data which was reflect the patient in his/her own) will be shared to other researchers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: April 2021- August 2021
Access Criteria: All applications related to scientific goals would be accepted.